CLINICAL TRIAL: NCT04876677
Title: Open Label, Prospective Study to Evaluate the Effect of Step-up From Non-extra Fine Inhaled Corticosteroids/Long Acting Beta2 Agonist (ICS/LABA) Dry Powder Inhaler (DPI) to Extra Fine Triple Therapy With CHF5993 DPI on Airway Geometry and Lung Ventilation Using Functional Respiratory Imaging (FRI) in Subjects With Advanced Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Functional Respiratory Imaging Study
Acronym: DARWiIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-05993BA1-08
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHF5993 (Experimental): Beclometasone Dipropionate (BDP) 100 μg/inhalation + Formoterol Fumarate (FF) 6 μg/inhalation + Glycopyrronium Bromide (GB) 12.5 µg/inhalation
  Interventions: Drug: Beclomethasone dipropionate/Formoterol Fumarate/Glycopyrronium

INTERVENTIONS:
Drug: Beclomethasone dipropionate/Formoterol Fumarate/Glycopyrronium — Two inhalations bid: 4 inhalations; total daily dose of 400/24/50 μg BDP/FF/GB

SUMMARY:
The purpose of this study is to evaluate the stepping-up effect from a double ICS/LABA DPI therapy to a triple DPI therapy on airway geometry and lung ventilation

ELIGIBILITY:
Inclusion Criteria:

1. Subject's signed Informed Consent Form;
2. Male or female ≥ 40 years of age;
3. Current smokers or ex-smokers of at least 10 pack-years,
4. Established diagnosis of COPD
5. Post-BD Forced Expiratory Volume in one second/Forced Vital Capacity (FEV1/FVC) < 0.7 and FEV1 ≤ 60% of predicted at V1
6. On a stable dose any non-extra fine ICS/LABA DPI twice daily regimen for at least 8 weeks before screening;
7. Presence of lung hyperinflation
8. Symptomatic subjects with COPD assessment test (CAT) score ≥ 10;
9. Documented history of ≥ 1 moderate or severe COPD exacerbation in the previous 12 months

Exclusion Criteria:

1. Pregnant or lactating woman;
2. Exacerbations defined as a sustained and acute deterioration of subject's symptoms and signs 30 days before screening;
3. A current asthma diagnosis;
4. Respiratory disorders other than COPD:
5. Cardiovascular diseases;
6. Evidence or history of other concurrent disease such as but not limited to hyperthyroidism, diabetes mellitus or other endocrine disease;
7. Medical history or current diagnosis of narrow-angle glaucoma;
8. History of lung transplant or lung reduction surgery;
9. ECG criteria: any clinically significant abnormal 12-lead ECG that in the investigator's opinion would affect efficacy or safety evaluation or place the subjects at risk;
10. Laboratory abnormalities;
11. Alcohol/drug abuse;
12. Contra-indications to Investigational medical products (IMPs), based on investigator judgement;
13. Documented Covid-19 diagnosis or its complications which have not resolved within 14 days prior to screening;

15. Positive molecular Covid-19 test within the last 72 hours before the remaining of screening activities.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
specific airway volume (siVaw) upon inspiration | change from baseline at 6 weeks
  CT-based airway volumes
specific airway resistance (siRaw) upon inspiration | change from baseline at 6 weeks
  CT-based airway volumes

SECONDARY OUTCOMES:
siVaw upon expiration | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
siRaw upon expiration | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
ventilation mapping | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
perfusion mapping | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
airway wall thickness upon inspiration | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
imaged lobe and lung volumes at Total Lung Capacity (TLC) and Functional Residual Capacity (FRC) | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
air trapping | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
low attenuation score at TLC | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
Percentile 15th at TLC | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography
regional lung deposition | change from baseline at 6 weeks
  calculated using Multidetector Computed Tomography

CONTACTS AND LOCATIONS:
Locations (8):
- Belgium (5):
  - OLV Hospital Aalst, Aalst
  - Centre medical Erpent - Residence, Erpent
  - AZ Zeno Knokke-Heist, Knokke
  - Heilige Familie AZ, Reet
  - AZ Delta, Roeselare
- Hungary (3):
  - Dr. Kenessey Albert Hospital, Balassagyarmat
  - National Koranyi Institute for TB and Pulmonology, Budapest
  - CRU Hungary Ltd, Miskolc

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Skloot GS, Guasconi A, Lavon BR, Georges G, De Backer W, Galkin D, Cortellini M, Panni I, Bates JHT. The effect of inhaled extrafine beclometasone dipropionate/formoterol fumarate/glycopyrronium bromide on distal and central airway indices, assessed using Functional Respiratory Imaging in COPD (DARWiIN). Respir Res. 2023 Oct 6;24(1):244. doi: 10.1186/s12931-023-02549-5. PMID 37803368